CLINICAL TRIAL: NCT04407104
Title: Allergy to Almond in Children: Diagnostic Values and Severity
Brief Title: Allergy to Almond in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI100
Record Dates: First submitted 2020-05-25; First posted 2020-05-29 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-05

CONDITIONS: Food Allergy in Children
Keywords: almond; tree nuts; atopy; allergy; children
MeSH Terms: conditions — Hypersensitivity | interventions — Patch Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: skin prick-test — retrospective study on data already collected
  Other Names: specific IgE; oral food challenge

SUMMARY:
Allergy to tree nuts are frequent in children but allergy to almond is one of the less described tree nuts allergy. The main objective of our study is to determine diagnostic values of skin prick-tests and specific IgE to almond in a population of children sensitized to almond and challenged in our unit from november 2013 to march 2020.

DETAILED DESCRIPTION:
Secondary objectives are

* description of allergic reactions to almond (symptoms, severity)
* modelisation of eliciting dose to almond in our population
* evaluation of the association between atopic comorbidities and allergy to almond in children sensitized to almond
* evaluation of the association between allergy to almond and the importance of skin and sIgE sensitization

ELIGIBILITY:
Inclusion Criteria:

* oral food challenge to almond performed in the pediatric allergy department of the University Hospital of Nancy from november 2013 and march 2020

Exclusion Criteria:

* doubtful or incomplete oral food challenge to almond

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children sensitized to almond and challenged in our unit
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-07-20 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-09-07 (Estimated)

PRIMARY OUTCOMES:
diagnostic values of skin prick-test and sIgE to almond | BASELINE

SECONDARY OUTCOMES:
allergic reactions during oral food challenge | BASELINE
  symptoms and severity
eliciting doses to almond | BASELINE
  ED05, ED10 and ED50
atopic comorbidities | BASELINE
  respiratory allergies, other food allergies, asthma

IPD SHARING:
Plan to Share IPD: No